CLINICAL TRIAL: NCT03032627
Title: Identifying Targets of Maladaptive Metabolic Responses in Heart Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Florida Hospital Cardiovascular Institute (Unknown); Sanford-Burnham Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMDFH 936207
Record Dates: First submitted 2017-01-17; First posted 2017-01-26 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac surgery (Other): Subjects will be recruited by a coordinator through electronic medical record (EMR) searches to identify those undergoing left ventricle assist device (LVAD) implantation and explantation, heart transplant, valve replacement or repair, endomyocardial biopsy during catheterization, and arterial bypass surgery. Prior to the procedure, potential subjects will be informed about the clinical study and if interested, they will be consented.
  Interventions: Procedure: Collection of discarded heart tissue

INTERVENTIONS:
Procedure: Collection of discarded heart tissue — Discarded heart tissue will be collected from patients undergoing the aforementioned cardiac surgeries.

SUMMARY:
The purpose of the research is to help researchers understand changes in metabolism in patients that develop heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are capable of giving informed consent.
2. Age 19-89
3. Diagnosis of chronic heart failure
4. Any patients scheduled for at least one of the following procedures:

   1. LVAD implantation or as recipient for cardiac transplantation.
   2. LVAD placement both as bridge to transplant and as destination therapy.
   3. LVAD explantation
   4. Valve replacement or repair
   5. Catheterization and myocardial biopsy for idiopathic cardiomyopathy
   6. Coronary artery bypass graft (CABG)

Exclusion Criteria:

1. Life expectancy less than 2 weeks
2. Diagnosed with following co-morbidities: cancer, chronic kidney disease (GFR≤30 or serum creatinine >2.1), active infection or treatment with antibiotics or persistent infectious disease (hepatitis, HIV, etc), cirrhosis, active substance abuse and/or alcohol dependence (≥ 14 alcoholic beverages per week).

Control Myocardial Tissue from Donor Hearts Inclusion Criteria

1. Samples collected from non-failing hearts deemed unsuitable for transplantation by TransLife because of either acute recipient issues or post-harvest evidence of pathology or positive but benign serology.
2. Normal cardiac function from medical records

Exclusion Criteria:

1. Pathological remodeling and extensive infarction with limited non-pathological regions of myocardium.
2. Abnormal or impaired cardiac function from medical records, which are self determinants for rejection as a donor organ.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Analyses of collected tissues | Restricted to the time around surgical procedure
  Tissue samples collected during surgery will be analyzed by way of immunoblot and qrtPCR of mRNA for metabolic enzymes on neutralized acid extracts.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Pratley, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braunwald E. Heart failure. JACC Heart Fail. 2013 Feb;1(1):1-20. doi: 10.1016/j.jchf.2012.10.002. Epub 2013 Feb 4. PMID 24621794
- [Background] Franklyn JA. The molecular mechanisms of thyroid hormone action. Baillieres Clin Endocrinol Metab. 1988 Nov;2(4):891-909. doi: 10.1016/s0950-351x(88)80023-5. No abstract available. PMID 2908318
- [Background] Grosjean O, Bluemenstock D. [Pulmonary and renal transplantations in the dog treated by single and later repeated neonatal injections of bone marrow]. C R Seances Soc Biol Fil. 1967 Sep;161(3):733-7. No abstract available. French. PMID 4229424
- [Background] Heath DF. Subcellular aspects of the response to trauma. Br Med Bull. 1985 Jul;41(3):240-5. doi: 10.1093/oxfordjournals.bmb.a072057. No abstract available. PMID 3896379
- [Background] Ingwall JS, Weiss RG. Is the failing heart energy starved? On using chemical energy to support cardiac function. Circ Res. 2004 Jul 23;95(2):135-45. doi: 10.1161/01.RES.0000137170.41939.d9. PMID 15271865
- [Background] Suyama K, Goldstein J, Aebersold R, Kent S. Regarding the size of Rh proteins. Blood. 1991 Jan 15;77(2):411. No abstract available. PMID 1898705
- [Background] Blahos J, Mertl L, Gregor O, Kotas J, Reisenauer R. [Stimulating effect of hypercalcaemia on basal gastric secretion (author's transl)]. Cas Lek Cesk. 1974 Aug 2;113(31):944-7. No abstract available. Czech. PMID 4410983
- [Background] Bucci E, Mignogna MD. [Diagnosis and prevention of stress in dental patients]. Dent Cadmos. 1986 May 31;54(9):77-8, 80, 82. No abstract available. Italian. PMID 3464497
- [Background] Torok B. Microcomputer-based recording system for clinical electrophysiology. Doc Ophthalmol. 1990 Sep;75(2):189-97. doi: 10.1007/BF00146555. PMID 2276319
- [Background] Polak J, Kotrc M, Wedellova Z, Jabor A, Malek I, Kautzner J, Kazdova L, Melenovsky V. Lipolytic effects of B-type natriuretic peptide 1-32 in adipose tissue of heart failure patients compared with healthy controls. J Am Coll Cardiol. 2011 Sep 6;58(11):1119-25. doi: 10.1016/j.jacc.2011.05.042. PMID 21884948
- [Background] Collins S. A heart-adipose tissue connection in the regulation of energy metabolism. Nat Rev Endocrinol. 2014 Mar;10(3):157-63. doi: 10.1038/nrendo.2013.234. Epub 2013 Dec 3. PMID 24296515
- [Background] Kovacova Z, Tharp WG, Liu D, Wei W, Xie H, Collins S, Pratley RE. Adipose tissue natriuretic peptide receptor expression is related to insulin sensitivity in obesity and diabetes. Obesity (Silver Spring). 2016 Apr;24(4):820-8. doi: 10.1002/oby.21418. Epub 2016 Feb 17. PMID 26887289